CLINICAL TRIAL: NCT04580082
Title: ADHOC Mindfulness-Based Research - An Intervention to Address Loneliness Among Older People Living With HIV
Brief Title: ADHOC Mindfulness-Based Research
Acronym: AMBR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mazonson & Santas Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20017 - 01D
Record Dates: First submitted 2020-09-28; First posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Hiv; Loneliness; Depression; Anxiety
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness lessons (Experimental): There are 14 lessons in total, each lasting approximately 20 minutes. Participants will be asked to listen to one lesson per day for 14 consecutive days, but to allow for possible missed days, they will have up to 25 days to complete as many of these 14 lessons as they can. The lessons will be delivered via the internet, and participants can use a variety of devices (e.g. smartphone, desktop computer, laptop computer, tablet) to access them. While the lessons cannot be downloaded, they are available for streaming anytime and anywhere there is an internet connection. Participants are welcome to revisit any lesson they have listened to previously, but are not allowed to "skip ahead" to other lessons until they have completed all preceding lessons. This is done because the lessons build on one another, which means that skipping lessons makes continued participation difficult. We will be able to track each participant's usage pattern and will analyze differences across users.
  Interventions: Behavioral: Mindfulness lessons
- Delayed-start Mindfulness Lessons (Other): The control group will not receive the intervention until the intervention group has completed lesson listening. During this waiting period, they will receive periodic emails letting them know that their turn to listen to lessons is coming soon.
  Once available, the control group will have 25 days to listen to the 14 lessons.
  Interventions: Behavioral: Mindfulness lessons

INTERVENTIONS:
Behavioral: Mindfulness lessons — 14 lessons on mindfulness, each lasting approximately 20 minutes.

SUMMARY:
The AMBR Study (ADHOC Mindfulness-Based Research Study) is a randomized controlled trial that examines the effectiveness of teaching mindfulness-based techniques through online lessons to combat loneliness, anxiety, and depression among people living with HIV over the age of 50. It is a substudy of the ADHOC study (ClinicalTrials.gov identifier NCT04311554).

DETAILED DESCRIPTION:
The AMBR Study is a randomized controlled trial that examines the effectiveness of teaching mindfulness-based techniques through online lessons to combat loneliness, anxiety, and depression among people living with HIV who are over the age of 50 and enrolled in ADHOC (ClinicalTrials.gov identifier NCT04311554). The intervention consists of 14 mindfulness audio lessons, each approximately 20-minutes long. The mindfulness lessons are designed to develop three core skills: concentration (the ability to maintain focus on present-moment experiences), clarity (the ability to pinpoint exactly what you are experiencing in each moment), and equanimity (openness to experience).

ELIGIBILITY:
Inclusion Criteria:

* ADHOC participant with a score of 4 or higher on the 3-item Loneliness Questionnaire from their ADHOC profile
* Clinical diagnosis of HIV
* Able to read and write in English
* Able and willing to provide online informed consent and complete study activities online
* Access to a smartphone or computer

Exclusion Criteria:

- Acute medical problem(s) requiring immediate inpatient treatment

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2020-05-21 (Actual); Primary Completion 2020-09-04 (Actual); Study Completion 2020-09-28 (Actual)

PRIMARY OUTCOMES:
Loneliness | Baseline and follow-up, 25 days
  Change in loneliness using the 3-Item Loneliness Questionnaire (3IL). 3IL scores range from 3-9, with higher scores indicating greater loneliness.

SECONDARY OUTCOMES:
Anxiety | Baseline and follow-up, 25 days
  Change in anxiety using the 7-item Generalized Anxiety scale (GAD-7). GAD-7 scores range from 0-21, with higher scores indicating more anxiety.
Depression | Baseline and follow-up, 25 days
  Change in depression using the 10-item Center for Epidemiologic Studies Depression scale (CES-D-10). CES-D-10 scores range from 0-30, with higher scores indicating more depression.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Mazonson, MD, MBA, Principal Investigator — Mazonson & Santas Inc.
Locations (1):
- Mazonson & Santas Inc, Larkspur, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Berko J, Mazonson P, Short D, Karris M, Ehui L, Gutner CA, Spinelli F, Zolopa A. Waitlist-controlled trial of an online intervention to address mental health among older people living with HIV. Antivir Ther. 2023 Dec;28(6):13596535231216311. doi: 10.1177/13596535231216311. PMID 38031911